CLINICAL TRIAL: NCT00003453
Title: Phase II Study of Antineoplastons A10 and AS2-1 In Patients With Carcinoma of the Adrenal Gland
Brief Title: Antineoplaston Therapy in Treating Patients With Stage IV Adrenal Gland Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Burzynski Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066485; BC-AD-02 (Other: Burzynski Research Institute)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2018-05-09 (Actual); Last update posted 2018-05-09 (Actual); Status verified 2018-04

CONDITIONS: Stage IV Adrenocortical Carcinoma
Keywords: recurrent adrenocortical carcinoma
MeSH Terms: conditions — Adrenocortical Carcinoma | interventions — antineoplaston A10; antineoplaston AS 2-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Antineoplaston therapy (Experimental): Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Interventions: Drug: Antineoplaston therapy (Atengenal + Astugenal)

INTERVENTIONS:
Drug: Antineoplaston therapy (Atengenal + Astugenal) — Patients with Stage IV Adrenal Gland Cancer will receive Antineoplaston therapy (Atengenal + Astugenal).
  The daily doses of A10 and AS2-1 are divided into six infusions, which are given at 4-hourly intervals. Each infusion starts with infusion of A10 and is immediately followed by infusion of AS2-1.
  Other Names: A10 (Atengenal); AS2-1 (Astugenal)ANP

SUMMARY:
Current therapies for Stage IV adrenal gland cancer provide very limited benefit to the patient. The anti-cancer properties of Antineoplaston therapy suggest that it may prove beneficial in the treatment of Stage IV adrenal gland cancer

PURPOSE: This study is being performed to determine the effects (good and bad) that Antineoplaston therapy has on patients with Stage IV adrenal gland cancer.

DETAILED DESCRIPTION:
OVERVIEW: This is a single arm, open-label study in which patients with Stage IV adrenal gland cancer receive gradually escalating doses of intravenous Antineoplaston therapy (Atengenal + Astugenal) until the maximum tolerated dose is reached. Treatment continues up to12 months in the absence of disease progression or unacceptable toxicity.

OBJECTIVES:

* To determine the efficacy of Antineoplaston therapy in patients with Stage IV adrenal gland cancer, as measured by an objective response to therapy (complete response, partial response or stable disease).
* To determine the safety and tolerance of Antineoplaston therapy in patients with Stage IV adrenal gland cancer.
* To determine objective response, tumor size is measured utilizing MRI scans, which are performed every 8 weeks for the first two years, every 3 months for the third and fourth years, every 6 months for the 5th and sixth years, and annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IV adrenal gland carcinoma that is unlikely to respond to existing therapy and for which no curative therapy exists
* Measurable disease by MRI or CT scan
* Tumor must be greater than 2 cm at the largest diameter for the lymph nodes located in the head, neck, axillary, inguinal, or femoral areas and at least 0.5 cm in the largest diameter for other localizations

PATIENT CHARACTERISTICS:

Age:

* 6 months and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 2 months

Hematopoietic:

* WBC at least 2,000/mm^3
* Platelet count at least 50,000/mm^3

Hepatic:

* Bilirubin no greater than 2.5 mg/dL
* SGOT/SGPT no greater than 5 times upper limit of normal
* No hepatic failure

Renal:

* Creatinine no greater than 2.5 mg/dL
* No history of renal conditions that contraindicate high dosages of sodium

Cardiovascular:

* No severe heart disease
* No uncontrolled hypertension
* No history of congestive heart failure
* No history of other cardiovascular conditions that contraindicate high dosages of sodium

Pulmonary:

* No severe lung disease

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 4 weeks after study participation
* No serious active infections or fever
* No other concurrent serious disease

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy and recovered
* No concurrent immunomodulating agents

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas) and recovered
* No concurrent antineoplastic agents

Endocrine therapy:

* Concurrent corticosteroids allowed

Radiotherapy:

* At least 8 weeks since prior radiotherapy and recovered

Surgery:

* Recovered from any prior operative procedure

Other:

* No prior antineoplaston therapy
* Prior cytodifferentiating agent allowed

Ages: 6 Months to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 1996-08-21; Primary Completion 2011-07-05 (Actual); Study Completion 2011-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Principal Investigator — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Burzynski Research Institute — http://www.burzynskiresearch.com
- See also: Burzynski Clinic — http://www.burzynskiclinic.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Six patients were recruited between August 1996 and February 2007. All study subjects were seen at the Burzynski Clinic in Houston, TX
Period: Overall Study
Arm/Group | Antineoplaston Therapy
Started | 6
Completed | 5 (One patient was not evaluable)
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 45.0 [0.67 to 64.75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response
Description: Objective response rate per Response Assessment in Neuro-Oncology (RANO) for target lesions and assessed by MRI: Complete Response (CR), disappearance of all disease sustained for at least four weeks; Partial Response (PR), >=50% decrease in the sum of the products of of the greatest perpendicular diameters of all measurable enhancing lesions, sustained for at least four weeks.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 5
Participants
  Complete Response | 1
  Partial Response | 1
  Stable Disease | 1
  Progressive Disease | 2

2. Secondary Outcome: Percentage of Participants Who Survived
Description: 6 months, 12 months, 24 months, 36 months, 48 months, 60 months overall survival
Time Frame: 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
Measure: Number; unit: Percentage of participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 6
Percentage of participants
  6 months overall survival | 83.3
  12 months overall survival | 66.7
  24 months overall survival | 50.0
  36 months overall survival | 33.3
  48 months overall survival | 33.3
  60 months overaall survival | 33.3

ADVERSE EVENTS:
Time Frame: 13 years, 5 months
Description: Adverse event data was collected through regular patient assessment and regular laboratory testing
Arm/Group | Antineoplaston Therapy
Serious Adverse Events (participants affected / at risk) | 4/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=6)
Ascites (non-malignant) (Gastrointestinal disorders) | 1 — The Ascites (non-malignant) was not related to Antineoplaston Therapy
Musculoskeletal/Soft Tissue - Other (Muscle Spasms) (Musculoskeletal and connective tissue disorders) | 1 — The Musculoskeletal/Soft Tissue - Other (Muscle Spasms) was not related to Antineoplaston Therapy
Fever (General disorders) | 1 — The Fever was not related to Antineoplaston Therapy.
Central Venous Catheter Infection (General disorders) | 1 — The Central Venous Catheter Infection was not related to Antineoplaston Therapy
Somnolence/depressed level of consciousness (Nervous system disorders) | 1 — The Somnolence/depressed level of consciousness was not related to Antineoplaston Therapy
Dizziness (Nervous system disorders) | 1 — The Dizziness was not related to Antineoplaston Therapy
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=6)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1
Allergic rhinitis (including sneezing, nasal stuffiness (Immune system disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 4
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 2
Lymphopenia (Blood and lymphatic system disorders) | 2
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 2
Platelets (Blood and lymphatic system disorders) | 2
Cardiac Arrhythmia - Other (Cardiac disorders) | 2
Hypertension (Cardiac disorders) | 3
Central venous catheter infection (General disorders) | 2
Non-functional central venous catheter (General disorders) | 2
Central venous catheter - Other (General disorders) | 2
Pain: Central venous catheter (General disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 5
Fever (General disorders) | 3
Insomnia (General disorders) | 1
Rigors/chills (General disorders) | 2
Sweating (diaphoresis) (General disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1
Edema/Fluid retention (General disorders) | 2
Anorexia (Gastrointestinal disorders) | 1
Ascites (non-malignant) (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Dental: teeth (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 2
Enteritis (inflammation of the small bowel) (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 4
Hemorrhage, GU: Bladder (Renal and urinary disorders) | 2
Infection - Other (Infections and infestations) | 1
Infection (documented clinically): Bladder (urinary) (Infections and infestations) | 1
Infection (documented clinically): Bronchus (Infections and infestations) | 1
Infection (documented clinically): Dental-tooth (Infections and infestations) | 1
Infection (documented clinically): Mucosa (Infections and infestations) | 1
Infection (documented clinically): Upper airway NOS (Infections and infestations) | 1
Infection with normal ANC: Abdomen NOS (Infections and infestations) | 1
Albumin, serum-low (hypoalbuminemia) (Investigations) | 3
Alkaline phosphatase (Investigations) | 4
Bicarbonate, serum-low (Investigations) | 2
Hypercalcemia (Investigations) | 1
Hypercholesteremia (Investigations) | 2
Hyperglycemia (Investigations) | 1
Hyperkalemia (Investigations) | 1
Hypernatremia (Investigations) | 3
Hypertriglyceridemia (Investigations) | 2
Hypocalcemia (Investigations) | 3
Hypoglycemia (Investigations) | 4
Hypokalemia (Investigations) | 6
Hypomagnesemia (Investigations) | 1
Hypophosphatemia (Investigations) | 2
Proteinuria (Investigations) | 2
SGOT (Investigations) | 3
SGPT (Investigations) | 1
Uric acid, serum-high (hyperuricemia) (Investigations) | 2
Musculoskeletal/Soft Tissue - Other (Muscle Spasms) (Musculoskeletal and connective tissue disorders) | 1
Confusion (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Mood alteration (Nervous system disorders) | 1
Mood alteration: Agitation (Nervous system disorders) | 1
Somnolence/depressed level of consciousness (Nervous system disorders) | 3
Pain: Abdomen NOS (Gastrointestinal disorders) | 4
Pain: Bladder (Renal and urinary disorders) | 1
Pain: Chest/thorax NOS (Musculoskeletal and connective tissue disorders) | 1
Pain: Head/headache (Nervous system disorders) | 3
Pain: Joint (Musculoskeletal and connective tissue disorders) | 1
Pain: Muscle (Musculoskeletal and connective tissue disorders) | 2
Pain: Neck (Musculoskeletal and connective tissue disorders) | 1
Pain: Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Renal/Genitourinary - Other (Renal and urinary disorders) | 1
Urinary frequency/urgency (Renal and urinary disorders) | 1
Flu-like syndrome (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No